CLINICAL TRIAL: NCT02202200
Title: An Open Label Multicenter, Phase I-II Study With Tumor Molecular Pharmacodynamic (MPD) Evaluation and Pharmacokinetics of PD-0332991 in Patients Suffering Metastatic Melanoma With BRAFv600 Mutated and CDKN2A Loss and Expression of Rb and Treated by Vemurafenib
Brief Title: Phase I-II Study With Tumor Molecular Pharmacodynamic (MPD) Evaluation and Pharmacokinetics of PD-0332991 in Patients Suffering Metastatic Melanoma
Acronym: OPTIMUM
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D20121106
Record Dates: First submitted 2014-07-25; First posted 2014-07-28 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Melanoma BRAF V600E/K Mutated; CDNKN2A Loss Defined
Keywords: Melanoma; BRAF mutated
MeSH Terms: conditions — Melanoma | interventions — palbociclib

ARMS (1):
- PD-0332991 (Experimental)
  Interventions: Drug: PD- 0332991

INTERVENTIONS:
Drug: PD- 0332991 — PD-0332991 Inhibitor of cyclin-dependant kinase (CDK) 8 schedules will be evaluated PD-0332991 PO QD either at 25 mg, 50 mg, 75 mg, 100 mg, 125 mg, 150 mg, 175 mg and 200 mg
  All patients will receive vemurafenib as background therapy ,bid at 720mg bid for the first group (during the first 2 cycle then 960 mg bid if good tolerance) and 960mg bid for all other patients

SUMMARY:
An open label multicentre, phase I-II study with tumour molecular pharmacodynamics (MPD) evaluation and pharmacokinetics of PD-0332991 added to vemurafenib in patients suffering metastatic melanoma with BR.

The main objective is to establish the Maximum Tolerated Dose (MTD) of PD-0332991 when added to standard vemurafenib therapy (960 mg BID). The estimated MTD is defined as the dose of PD-0332991 combined with vemurafenib that will be associated with a prespecified proportion of patients experiencing a Dose-Limiting Toxicity (DLT), ie, 1/3.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Stage IV or un-resectable stage III melanoma
* Presence of BRAF V600E/K mutation and CDNKN2A loss and expression of Rb using immunohistochemistry in a recent metastatic sample (< 6 months)
* A previous exposure to BRAF inhibitor or combination of BRAF and MEK inhibitors therapy is allowed unless it has been stopped more than 3 months before study enrolment(This will defined the two strata of the trial)
* No previous therapy by MEK inhibitor unless associated with BRAF inhibitors
* No previous therapy with the AKT/PI3K pathway inhibitor
* Patients should have a tumour available for repeated biopsies for pharmacodynamics evaluation
* Life expectancy of > 3 months
* ECOG performance status <2
* Signed informed consent
* Patient with health insurance coverage
* No patient under guardianship or curators

Exclusion Criteria:

* Inadequate hepatic function defined as serum bilirubin>25 μmol/l, transaminases > 3.0 times the upper limit of normal (ULN) or 5ULN in cases of liver metastases;
* Inadequate bone marrow function defined as absolute neutrophil count<1500/mcl, platelets<150000/mcl and haemoglobin<8g/dL
* Inadequate renal function with serum creatinine>2.0mg/dl) and /or creatinine clearance< 60 ml/min
* Untreated brain metastases : Patients with brain metastases will be eligible if they have completed treatment 1 months prior to the start of study medication, have discontinued corticosteroid treatment for these metastases for at least 5 days, and are neurologically asymptomatic
* Myocardial infarct or unstable angina within the past 6 months
* Concomitant take of drugs known to be strong inhibitor or inducers of CYP314
* HIV positive.
* Chemotherapy, immunotherapy within 4 weeks
* Drugs interfering with PD-0332991 and vemurafenib metabolism
* Malabsorption syndrome or other condition that would interfere with enteral absorption
* Congenital long QT syndrome or screening QTc > 470 msec
* Need for chronic corticosteroid therapy of ≥10 mg of prednisone per day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-11 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Occurrence within the first 2 cycles of treatment of a DLT | 42 Days
  DLTs, serious adverse events and adverse events leading to treatment discontinuations will be determined as follows:
  * Any grade 3 or more non-haematological toxicity excluding:
  * Grade 3 asymptomatic increase in liver function tests (AST, ALT, ALP) reversible within 7 days for subjects without liver involvement, or grade 4 for subjects with liver involvement.
  * Grade 3 vomiting if it is encountered despite adequate and optimal therapy (e.g. 5HT3 antagonists and corticosteroids).
  * Grade 3 diarrhoeas if encountered despite adequate and optimal anti diarrhoea therapy.
  * Confirmed grade 3 QTc prolongation (QTc >500 msec) that persists after correction of other possible causes such as electrolyte imbalance
  * Grade 4 hyperlipidemia if it is encountered despite adequate and optimal therapy.
  * Any grade 4 neutropenia of > 5 days duration, or febrile neutropenia lasting for more than 1 day.
  * Grade 4 thrombocytopenia > 1 day, or grade 3 with bleeding.

SECONDARY OUTCOMES:
Efficacy | 42 Days
  Occurrence of clinical benefit (defined as Complete Response (CR), Partial Response (PR) or stable disease (SD)) and progressive disease based on the best overall response which depends on the tumour evaluations assessed using RECIST at the end of each 2 cycles.
1 year survival rate | 1 year
  survival
Tolerance | 6 months
  Occurrence of clinically significant changes in a laboratory parameter and/or vital signs judged to be related to the trial medication within the first 6 months.

OTHER OUTCOMES:
Pharmacodynamic | 42 days
  * Changes from baseline of ANC and platelet levels
  * Efficiency on the cell-cycle machinery and proliferation (tumor sample)
  * Induction of senescence: will be evaluated using the senescence β-Galactosidase assay (Cell Signaling Technology)
  * Induction of apoptosis: will be performed using TUNEL staining with the ApopTag Peroxidase In Situ Apoptosis Detection Kit (Millipore).

CONTACTS AND LOCATIONS:
Locations (1):
- Saint-Louis Hospital, Paris, Paris, France

REFERENCES:
- [Derived] Louveau B, Resche-Rigon M, Lesimple T, Da Meda L, Pracht M, Baroudjian B, Delyon J, Amini-Adle M, Dutriaux C, Reger de Moura C, Sadoux A, Jouenne F, Ghrieb Z, Vilquin P, Bouton D, Tibi A, Huguet S, Rezai K, Battistella M, Mourah S, Lebbe C. Phase I-II Open-Label Multicenter Study of Palbociclib + Vemurafenib in BRAF V600MUT Metastatic Melanoma Patients: Uncovering CHEK2 as a Major Response Mechanism. Clin Cancer Res. 2021 Jul 15;27(14):3876-3883. doi: 10.1158/1078-0432.CCR-20-4050. Epub 2021 May 4. PMID 33947696